CLINICAL TRIAL: NCT02504437
Title: Therapy of Preconditioned Autologous BMMSCs for Patients With Ischemic Heart Disease
Acronym: TPAABPIHD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Academy Military Medical Science, China (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xuetao Pei, Director, Head of South China Research Center for Stem Cell & Regenerative Medicine, AMMS, Guangzhou, China., Academy Military Medical Science, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMMSC-1
Record Dates: First submitted 2015-07-14; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Myocardial Infarction; Acute Myocardial Infarction; Ischemic Cardiomyopathy
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- pre-conditioned BMMSCs (Experimental): autologous bone marrow mesenchymal stem cells (BMMSCs) with hypoxia pre-condition and endothelial pre-induction.
  Interventions: Biological: BMMSCs
- BMMSCs (Active Comparator): autologous bone marrow mesenchymal stem cells (BMMSCs) without pre-condition.
  Interventions: Biological: BMMSCs
- Controls (Sham Comparator): standard therapy without autologous bone marrow mesenchymal stem cells (BMMSCs) infusion.
  Interventions: Biological: BMMSCs

INTERVENTIONS:
Biological: BMMSCs

SUMMARY:
The purpose of the present study is to evaluate the efficacy of the preconditioned autologous bone marrow mesenchymal stem cells for patients with ischemic heart diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age under 75;
* Clinical diagnosis of acute Myocardial Infarction, chronic Myocardial Infarction and Ischemic Cardiomyopathy
* NYHA (New York Heart Association) grade: III-IV, LVEF (left ventricular ejection fraction): 25-50%;
* No infection diseases including HBV (hepatitis B virus), HCV (hepatitis C virus ), syphilis and AIDS;
* No psychiatric illnesses and speaking dysfunction;
* Informed consent.

Exclusion Criteria:

* More than 75 years old;
* LVEF<24%;
* Unstable hemodynamics, shock;
* Severe infection;
* Patients have tumor or other lethal diseases (expectation of life<6 months);
* Radiation patients;
* hematopoietic malignancy including Haemophiliacs;
* Anemia (Hb<100g/L);
* The other clinical trial participants within one month;
* Abnormal increasing of the blood biochemical indicators that is not explained by the conditions;
* Informed refusal.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
LVEF (left ventricular ejection fraction) | one year

REFERENCES:
- [Background] Gao LR, Pei XT, Ding QA, Chen Y, Zhang NK, Chen HY, Wang ZG, Wang YF, Zhu ZM, Li TC, Liu HL, Tong ZC, Yang Y, Nan X, Guo F, Shen JL, Shen YH, Zhang JJ, Fei YX, Xu HT, Wang LH, Tian HT, Liu DQ, Yang Y. A critical challenge: dosage-related efficacy and acute complication intracoronary injection of autologous bone marrow mesenchymal stem cells in acute myocardial infarction. Int J Cardiol. 2013 Oct 9;168(4):3191-9. doi: 10.1016/j.ijcard.2013.04.112. Epub 2013 May 4. PMID 23651816